CLINICAL TRIAL: NCT02323919
Title: Improving Long Term Exercise in Older Cardiac Patients
Brief Title: Long-term Exercise in Older Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Dr. Shirley Moore, Professor and Associate Dean, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL084767
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
Keywords: myocardial infarction; coronary artery bypass graft (CABG); angioplasty; exercise; cardiac patient; physical activity
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SystemCHANGE (Active Comparator): consists of self-efficacy enhancement and relapse prevention strategies, but is primarily anchored in a set of behavior change strategies based on System Improvement techniques.
  Interventions: Behavioral: CHANGE+
- CHANGE+ (Active Comparator): is based on several cognitive-behavioral theoretical frameworks: Social Problem-solving Model, Self-efficacy theory, Expectancy-value theory and Relapse Prevention theory.
  Interventions: Behavioral: SystemCHANGE
- Usual Care (Placebo Comparator): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: SystemCHANGE — consists of a series of five small-group (six to eight people) education sessions provided in three 1.5 -hour sessions once a week during the last three weeks of the CRP and in two sessions held at one and two months following completion of their CRP. An experienced cardiac nurse or exercise physiologist trained in the intervention protocol taught each of the sessions. In a series of structured activities, participants were taught to use behavior change strategies consistent with the respective intervention models. A series of three monthly booster calls were made during months four, five and six following the last intervention class and individuals were coached in the use of strategies consistent with the respective interventions.
  Arms: CHANGE+
Behavioral: CHANGE+ — consists of a series of five small-group (six to eight people) education sessions provided in three 1.5 -hour sessions once a week during the last three weeks of the CRP and in two sessions held at one and two months following completion of their CRP. An experienced cardiac nurse or exercise physiologist trained in the intervention protocol taught each of the sessions. In a series of structured activities, participants were taught to use behavior change strategies consistent with the respective intervention models. A series of three monthly booster calls were made during months four, five and six following the last intervention class and individuals were coached in the use of strategies consistent with the respective interventions.
  Arms: SystemCHANGE
Behavioral: Usual Care — Participants will receive only the routine care provided to CRP patients. This care consists of assessment of exercise capacity, graduated exercise training (consisting of exercising three times a week at the cardiac rehabilitation center on treadmill or cycle, counseling about safe exercise {warm-up procedures, pulse taking, attending to body cues for exertion levels} and advisement to exercise on days between CRP sessions). At the end of the CRP, individuals are given an exercise prescription that includes their target heart rate and they are counseled to exercise at least 5 times a week for 30 minutes. This information is provided by the CRP personnel, usually in the form of individual informal conversations during exercise at the CRP.
  Arms: Usual Care

SUMMARY:
Using a randomized clinical trial with 3 groups, the investigators will conduct a head-to-head evaluation of two different theoretically-based interventions, SystemCHANGE and CHANGE+, as compared to Usual Care to improve the adoption and maintenance of exercise in older cardiac patients. SystemCHANGE, a novel intervention that focuses on environmental change uses System Improvement strategies to increase exercise, will be compared to CHANGE+ (an intervention based contemporary cognitive behavioral strategies). Study questions are: (1) Is there a difference between SystemCHANGE, CHANGE+ and Usual Care in exercise adoption when controlling for covariates (age, race, functional capacity, body fat, co-morbidity, muscle or joint pain, exercise experience, home and neighborhood environment, and depression), for individuals following a cardiac rehabilitation program (CRP)? (2) Is there a difference between SystemCHANGE, CHANGE+, and Usual Care in exercise maintenance when controlling for covariates? (3) Do system changes, social support for exercise, problem-solving skills, motivation, health beliefs, and exercise self-efficacy mediate the effects of SystemCHANGE, CHANGE+, or Usual Care on exercise adoption? (4) Do system changes, social support for exercise, problem-solving skills, motivation, health beliefs, and exercise self-efficacy mediate the effects of SystemCHANGE, CHANGE+ and CHANGE+ interventions in terms of health care spending, labor force participation and earnings, and household productivity?

Older persons (N=420) recovering from cardiac events will be randomly assigned to the three groups. Measures of exercise adoption and maintenance (# of metabolic equivalents {METS} expended, and whether or not a subject remains exercising) will be taken for 1 year after completion of a CRP using heart rate wristwatch monitors, exercise diaries, and 7-Day Recall Survey. The effect of covariates also will be assessed. Mechanisms by which the interventions achieve their effects will be determined. Multivariate analyses will examine and compare the effects of the interventions over time. A cost-effectiveness analysis also will be conducted.

DETAILED DESCRIPTION:
Assisting individuals to adopt and maintain lifestyle exercise after a cardiac event remains challenging. The purpose of this 3-group, randomized controlled trial was to test two theoretically distinct behavior change interventions against a usual care (UC) group to increase lifestyle exercise after a cardiac event. In a new intervention, SystemCHANGE (SC), based on process improvement and ecological theories, participants were taught to use a series of small self-designed experiments to change their daily routines associated with exercise. The emphasis was on changing systems in their lives rather than relying on motivation or memory. The second intervention, CHANGE+ (C+), based on cognitive behavioral theory, included contemporary approaches to increase self-efficacy, motivation, and problem-solving skills.

Sample

The sample consisted of a convenience sample of 379 individuals who were consecutively recruited from five Phase II cardiac rehabilitation programs (CRP) in the greater Cleveland, Ohio area. Forty percent of the participants approached agreed to participate and were randomized. Of the 406 subjects consented, 379 completed the study. Subjects were randomly assigned to one of three study arms: SystemCHANGE (process improvement model program of health behavior change), CHANGE+ (cognitive behavioral model program of health behavior change), or Usual Care. All subjects had a recent cardiac event (myocardial infarction, coronary artery bypass surgery and/or percutaneous coronary intervention) and were participating in a Phase II cardiac rehabilitation program. Subjects were recruited near the end of their program and followed for one year after cardiac rehabilitation. Subjects were included if they were greater than 55 years of age and able to read and speak English; they were excluded if they met criteria for being at high risk for safe exercise participation following a cardiac event (ejection fraction < 30%, decrease in systolic blood pressure of > 15 mmHg with exercise, serious arrhythmias at rest or exercise induced, and exercise induced ischemia indicated by angina > 2 mm ST segment depression on the electrocardiogram).

Intervention Protocols

Both the CHANGE+ and SystemCHANGE interventions consist of a series of five small-group (six to eight people) education sessions provided in three 1.5-hour sessions once a week during the last three weeks of the CRP and in two sessions held at one and two months following completion of their CRP. An experienced cardiac nurse or exercise physiologist trained in the intervention protocol taught each of the sessions. In a series of structured activities, participants were taught to use behavior change strategies consistent with the respective intervention models. A series of three monthly booster calls were made during months four, five and six following the last intervention class and individuals were coached in the use of strategies consistent with the respective interventions. Usual Care consisted of only the routine care provided at the CRP. All participants received the usual CRP prescribed structured exercise and individual and group classes (four) on diet modification and stress reduction that are part of routine care at the CRPs. At the end of the CRP, all individuals were given an exercise prescription that included their target heart rate and counseled to exercise at least five times a week for 30 minutes.

Measures

Three dimensions of exercise were measured: frequency, amount, and maintenance. Exercise frequency was the number of sessions exercised (of at least 10 minutes duration) over a given period of time. Exercise amount was the number of hours exercised and reflected both the frequency and the duration of each exercise session. Exercise was measured using portable wristwatch heart rate monitors (Polar RS400) and exercise diaries. Data from the monitors was used as the primary data source with diary data used as backup if data from the monitor were not available (i.e., forgot to put on the monitor, monitor malfunction). The heart rate (HR) monitor memory was programmed to record HR at 5-second intervals during an exercise session. Standardized, validated measures were also obtained at baseline, two, six, and twelve months of: system changes, social support for exercise, problem-solving skills, motivation, health beliefs, and exercise self-efficacy. Measures were also obtained on possible moderating and confounding variables: age, race, functional capacity, body fat, co-morbidity, muscle or joint pain, exercise experience, home and neighborhood environment, and depression.

Procedures

Individuals who met study inclusion criteria were enrolled during the sixth to eighth week of the CRP and written informed consent was obtained. Baseline measures were obtained in a private interview at the CRP center. The intervention began week ten of the subjects' CRP. At the end of their CRP, subjects were given HR monitors and exercise diaries and were directed to return mail them during each of the next twelve months. The number of hours exercised during exercise adoption (months one through three) and maintenance (months four through twelve) was calculated. Multiple linear regression was used to determine if study group membership predicted exercise adoption and maintenance. Mediation analysis was also conducted.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years and older
* myocardial infarction
* CABG
* percutaneous transluminal coronary angiography (PTCA)
* completing a Phase II cardiac rehabilitation program
* all patients will be approved for the ability to safely perform exercise by the cardiac rehabilitation program prior to entrance into the study.

Exclusion Criteria:

* children
* non-English speaking
* current valve surgery
* presences of neurological deficits
* renal (acute renal failure) or pulmonary complications (pneumonia, severe congestive heart failure)
* obvious musculoskeletal functional disabilities
* patients displaying any of the following cardiac characteristics at the time of discharge from the hospital also will be excluded:

  1. severe left ventricular dysfunction (ejection fraction <20%)
  2. decrease in systolic blood pressure >15 mmHg with exercise
  3. serious arrhythmias at rest or exercise induced, and (4) exercise-induced ischemia indicated by angina> 2 mm of ST depression on the ECG, if they met criteria for being at high risk for safe exercise participation following a cardiac event.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Objectively measured hours of exercise/month | study months 1-13